CLINICAL TRIAL: NCT03276416
Title: RAPP-children, Rhinitis & Asthma in Patient Perspective: Development and Validation of a Questionnaire for Quality of Life Evaluation in Children With Asthma and Allergic Rhinitis
Acronym: RAPP
Status: Completed | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 7/2017_A
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 150 children with concomitant asthma and rhinitis: Baseline and one-month administration of RAPP-children, RHINASTHMA-children, C-ACT, VAS, Kiddy KINDLE, GRS. Baseline and one-month spirometry.

SUMMARY:
This observational study aims at developing and validating a simple questionnaire to be routinely applied in the clinical practice, for the evaluation of the quality of life in children with concomitant asthma and allergic rhinitis. The study consists of two phases:

Phase 1: Development of the RAPP-children questionnaire starting from the validated RHINASTHMA-children questionnaire.

Phase 2: Administration and validation of the RAPP-children questionnaire. 150 children with concomitant asthma and allergic rhinitis will be followed-up for one month. Both at baseline and after one month, the RAPP children and several other standardized questionnaires will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 11 years
* Concomitant asthma and allergic rhinitis
* Males and Females

Exclusion Criteria:

* Immunological and metabolic systemic disease
* Major malformations of the upper airways
* Active smoker

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A study population of 150 children with concomitant asthma and allergic rhinitis, aged 6 to 11 years, both males and females, followed-up for one month at the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (IBIM CNR).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
RAPP-children response patterns | 1 months
  Multivariate analyses of the responses to the RAPP-children questions

SECONDARY OUTCOMES:
RHINASTHMA-children response patterns | 1 months
  Frequency distributions of the responses to the RHINASTHMA-children
C-ACT response patterns | 1 months
  Frequency distributions of the responses to the C-ACT (Childhood Asthma Control Test)
VAS response pattern | 1 months
  Frequency distribution of the response to the VAS (Visual Analog Scale)
Kiddy-KINDL response patterns | 1 months
  Frequency distributions of the response to the Kiddy-KINDL
Pulmonary function: FEV1 | 1 months
  Forced expiratory volume in the first second
Pulmonary function: FVC | 1 months
  Forced vital capacity
Pulmonary function: FEF25-75 | 1 months
  Forced expiratory flow at 25-75%

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

REFERENCES:
- [Derived] Fasola S, Montalbano L, Ferrante G, Cilluffo G, Malizia V, Baiardini I, Braido F, Viegi G, La Grutta S. RAPP-children: A new tool for assessing quality of life in patients with asthma and rhinitis. Clin Exp Allergy. 2020 Jun;50(6):662-671. doi: 10.1111/cea.13599. Epub 2020 Mar 25. PMID 32163631